CLINICAL TRIAL: NCT03460548
Title: A Multicentre Randomized Trial Comparing the Efficacy and Safety of REMOGEN® Omega Versus Cationorm® in the Treatment of Patients Suffering From Dry Eye
Brief Title: REMOGEN® Omega Versus Cationorm® in the Treatment of Patients Suffering From Dry Eye
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOGA-CT-1501
Record Dates: First submitted 2018-02-28; First posted 2018-03-09 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remogen (Experimental)
  Interventions: Device: Remogen
- Cationorm (Active Comparator)
  Interventions: Device: Cationorm

INTERVENTIONS:
Device: Remogen — instil 1 drop of the product in each eye, 4 times per day
  Arms: Remogen
Device: Cationorm — instil 1 drop of the product in each eye, 4 times per day
  Arms: Cationorm

SUMMARY:
The efficacy and safety of Remogen® Omega in the treatment of dry eye signs and symptoms will be investigated in comparison to Cationorm®.

ELIGIBILITY:
Inclusion Criteria:

* With at least a 3-month documented history of bilateral dry eye
* With a score of ocular surface staining with fluorescein (OSSF) ≥ 4 and ≤ 9 on the Oxford scale
* With at least one objective sign of tear deficiency
* With Ocular Surface Disease Index (OSDI) score of ≥ 18

Exclusion Criteria:

* Refractive surgery within 12 months prior to selection
* Any other ocular surgery or ocular trauma within 6 months prior to selection
* Systemic or local use of one of the following medications: glucocorticosteroids, cyclosporine A, antibiotics, NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
OSSF | Day 28
  Ocular surface staining with fluorescein (OSSF)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, MD, PhD, Principal Investigator — Quinze-Vingts Hospital, Paris, France
Locations (1):
- Quinze-Vingts Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No